CLINICAL TRIAL: NCT04461860
Title: Assessment of Pain of Pelvic Congestion Syndrome Treated by Coils Embolization (SCVPC)
Brief Title: Assessment of Pain of Pelvic Congestion Syndrome Treated by Coils Embolization
Acronym: SCVPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SCVPC (29BRC20.0089)
Record Dates: First submitted 2020-06-19; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-05

CONDITIONS: Pelvic Pain
Keywords: syndrome; pain; pelvic; vein; embolization
MeSH Terms: conditions — Pelvic Pain; Syndrome; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Summary:

Main Objective: to evaluate the efficacy of pelvic gonadal vein embolization with coils in treatment of pelvic congestion syndrome Methods: retrospective study included 25 patients in the University hospital of Brest.

The Primary Outcome Measure: To evaluate (to measure) pain relief using visual analogous scale (VAS) before and after gonadal vein embolization for pelvic congestion syndrome The Secondary Outcome Measures were to assess the impact of the treatment on specific and general symptoms through a survey.

DETAILED DESCRIPTION:
A retrospective, non-invasive monocentric study of our Hospital 10-year registry (including data on MRI angiography and Vascular Doppler Ultrasound) of patients who have already undergone coil embolization of pelvic gonadal vein in treatment of pelvic congestion syndrome. These patients will be contacted by phone to participate in the study. An information letter will be handed out and the study protocol will be explained to the patients. After obtaining their written consent, they will be asked to fill out the study's validated questionnaire at home and return it to us through pre-paid regular mail. A face to face interview with the patient will be scheduled to assess the correlation between patient's clinical symptoms and survey results. There will be no change in patient's routine follow-up care.

All physician investigators of the study are experts in their field of medicine (e.g. interventional MRI angiography, vascular disease).

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of pelvic congestion syndrome documented by Vascular Doppler ultrasound and vascular dynamic MRI
* Failed medical treatment.
* > 18 years < 60 years old

Exclusion Criteria:

* < 18 years old
* Under legal guardian
* Asymptomatic pelvic congestion syndrome
* Psychiatric disorder
* Endometriosis.
* Chronic pelvic disease
* Pregnancy
* Neoplasia
* Acute intermittent porphyria

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: women > 18 years old with at least 1 previous pregnancy and delivery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Pelvic congestion pain relief | pre-embolization and 1 month post-gonadal vein embolization
  To evaluate (to measure) pain relief using visual analogous scale before and after gonadal vein embolization for pelvic congestion syndrome. A high score means a worse outcome.

SECONDARY OUTCOMES:
evaluation of specific pelvic syndrome symptoms using a self-reported questionnaire survey | pre-embolization and 1 month post-gonadal vein embolization
  to assess the impact of gonadal vein embolization on specific symptoms of pelvic congestion syndrome through a self-reported questionnaire survey.
evaluation of general pelvic syndrome symptoms using a self-reported questionnaire survey | pre-embolization and 1 month post-gonadal vein embolization
  to assess the impact of gonadal vein embolization on general symptoms of pelvic congestion syndrome through a self-reported questionnaire survey.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the end of the study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.